CLINICAL TRIAL: NCT03372824
Title: Oral Glucose Tolerance Test (OGTT), HbA1c or Glycated Albumin - Can we Reduce the Need for OGTT in Pregnancy?
Brief Title: Glycated Albumin in Pregnancy
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUS-ID651
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2017-12

CONDITIONS: Gestational Diabetes
Keywords: mass screening
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Primiparas above 25 years of age, singleton pregnancy

SUMMARY:
This is an observational study at the Obstetrical outpatient clinic at Stavanger University Hospital, Norway. The purpose of the study is to compare glycated albumin and glycated hemoglobin (HbA1c), both markers of "long-term blood sugar" with oral glucose tolerance test (OGTT). The OGTT is a screening test for gestational diabetes, a condition that increases risk of adverse pregnancy outcome for mother and child. The risks are reduced with good glycaemic control throughout pregnancy, therefore, it is important to screen for gestational diabetes.

DETAILED DESCRIPTION:
According to the new guideline by the Norwegian Directorate of Health published april 2017, screening for gestational diabetes is increased. All pregnant women with a slight risk, approximately 70 % of pregnant women i Norway, should have an OGTT performed in gestational week 24-28. Among those women, all primiparas above the age of 25 years old.

The investigators will include 150 primiparas above the age of 25 years old in the study. The women will be asked to participate in the study when they attend an ultrasound examination at the Obstetric outpatient clinic in gestational week 18-20. Prior to inclusion, participants need to sign written informed consent.

Included women will get an appointment for OGTT in gestational week 24-28 at the Clinical trial unit, Stavanger University hospital. The OGTT will be performed according to national guidelines. The participants will fill in a single questionaire with information on age, height, ethnicity, whether there is diabetes in close family, any other illnesses, smoking habits and other medications/supplements.

In addition, to blood sugar levels, markers of importance for glycaemic control, iron status and vitamin-D status will be analyzed.

Women diagnosed with gestational diabetes or overt diabetes mellitus, will be followed up according to national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* primiparas >25 years old
* singleton pregnancy

Exclusion criteria:

- prior diagnosed with diabetes

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primiparas above the age of 25 years old at conception. Women will be asked to participate in the study when they atttend an ultrasound examination at the Obstetrical outpatient clinic, Stavanger University Hospital, in gestational week 18-20.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Glycated albumin reference interval in pregnancy | gestational week 24-28
  Glycated albumin will be analyzed by a new method based on mass spectrometry. Glycated albumin will be analyzed in blood samples taken during the OGTT.

SECONDARY OUTCOMES:
Oral glucose tolerance test in pregnancy | Gestational week 24-28
  The oral glucose tolerance test (OGTT) will be performed according to national guidelines as a screening test for gestational diabetes
HbA1c | Gestational week 24-28
  HbA1c, long-term bloodsugar, will be analyzed in blood sample taken during the OGTT for all participants
Iron status | Gestational week 24-28
  Iron status might effect the HbA1c Level. We will analyse iron status in blood samples collected at the OGTT for all participants.
Glycaemic control | Gestational week 24-37
  For women diagnosed with gestational diabetes, we will register blood sugar measurements from diagnosis until gestational week 37. These measurements will be compared to HbA1c and glycated albumin levels in blood sample taken in gestational week 37
Preeclampsia | From gestational week 20 until 1 week postpartum
  Pregnancy outcome. New onset systolic blood pressure >140, diastolic blood pressure >90 after gestational week 20 and proteinuria 2+ according to urine dipstick, will be registered as preeclampsia
Induction of labour | At delivery
  Register pregnancy outcome. Induction of Labour and indication for induction will be registered.
APGAR | At delivery
  Register pregnancy outcome. APGAR score (Appearance, Pulse, Grimace, Activity, Respiration) of the newborn will be registered for 1 minute, 5 minute and 10 minutes after delivery.
Birth weight | At delivery
  Register pregnancy outcome. Birth weight (gram) of the newborn will be registered
Admission to neonatal intensive care unit | At delivery
  Register pregnancy outcome. Admission to neonatal intensive care unit will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Johanne H Toft, MD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No